CLINICAL TRIAL: NCT06528535
Title: Evaluation of a Health Promotion Intervention on Food Safety in Women During Pregnancy
Acronym: NPTM2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: NutriPouTiMoun2
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Food Safety; Pregnancy Related; Health Promotion
Keywords: French Guiana; Pregnancy; Food safety; Health promotion; Nutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, urine, serum, plasma, hair, placenta
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - intervention: Pregant women living in French Guiana who benefited from a health promotion intervention
  Interventions: Other: Health promotion intervention
- Group 2 - control: Pregant women living in French Guiana who did not benefit from a health promotion intervention

INTERVENTIONS:
Other: Health promotion intervention — Health promotion activities on nutrition with distribution of baskets of fresh fruits and vegetables
  Groups: Group 1 - intervention

SUMMARY:
This is a comparative, observational study aiming to compare the diversity of the diet during pregnancy of women who have benefited from a health promotion intervention and who have not

DETAILED DESCRIPTION:
In the Nutri Pou Ti'moun 1 project on food and nutritional insecurity during pregnancy, the inclusion of pregnant women began at the end of January 2023. As of 24 July 2023, 625 pregnant women had been included in the study. The main aim of this study is to estimate the prevalence of household food insecurity among pregnant women admitted for childbirth in one of Guyana's maternity units. Of the women included in this project, 13% were being monitored by one of French Guiana's mother and child protection centres (PMI).

In order to improve pregnancy monitoring for women and adapt to the specific characteristics of the region, the range of antenatal care services is diversified and complementary. For example, the PMI centres mainly monitor pregnant women who are not, or are no longer, entitled to social security benefits or who are affiliated to the State Medical Aid (AME) scheme, while the private sector mainly monitors women who are affiliated to one of the social security schemes. In the sub-group of women followed up by the PMI, the proportion of women in a precarious situation is therefore higher. In view of the issues raised by the Nutri Pou Ti'moun 1 project, it would seem appropriate to describe the situation of food and economic insecurity with greater statistical power in this sub-group of interest, and therefore to over-represent the women followed up by the PMI in the total sample.

The French Guiana Perinatal Network is one of the health networks defined by the law of 4 March 2002, relating to patients' rights and the quality of the health system, as follows: 'The purpose of health networks is to promote access to care, coordination, continuity or interdisciplinarity of health care provision, particularly that which is specific to certain populations, pathologies or health activities. They provide care tailored to the needs of the individual in terms of health education, prevention, diagnosis and care. They may take part in public health initiatives.

The French Guiana Perinatal Network is an association, created in 2002, whose main objective is to improve the quality of care and monitoring of pregnant women and newborn babies, as well as vulnerable children in French Guyana.

The French Guiana Perinatal Network implements a health promotion initiative on nutrition during pregnancy (between the 4th and 7th months) based on :

* Health mediation;
* Group workshops on nutrition, self-esteem, appropriate physical exercise, food budget management, breastfeeding and parenthood;
* Distribution of a basket of fresh fruit and vegetables

The patients benefiting from this intervention will be women attending one of the PMI centres taking part in the study.

These actions are likely to modify the prevalence of food insecurity among beneficiaries. Thus, it seems relevant :

* To identify, among the patients included, those who had benefited from this intervention in order to avoid introducing a bias when measuring the judgement criteria;
* To include patients followed up in the PMI centres of one of the participating centres and who had benefited from the intervention;
* To compare the prevalence of food insecurity between those who had benefited from the Réseau Périnat intervention and those who had not.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group : Pregant women living in French Guiana during their pregancy and who benefited from the intervention
* Control group : Pregant women living in French Guiana during their pregancy and who did not benefit from the intervention

Exclusion Criteria:

* Refusal to participate to the study
* No authorisation of participation from legal representatives for minor participants
* Participants under guardianship or trusteeship

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women living in French Guiana at the moment of the study, who have benefited or not from health promotion intervention on nutrition
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Description of diet during pregancy | At inclusion
  To describe the diet of pregnant women among women who benefited from the health promotion intervention and those who didn't from a questionnaire

SECONDARY OUTCOMES:
Prevalence of food insecurity | At inclusion
  To estimate food insecurity of pregnant women monitored in PMI using the Minimum Dietary Diversity for Women (MDD-W) score
Description of socio-demographic characteristics of participants | At inclusion
  To compare the socio-demographic characteristics of pregnant women who benefited from the intervention with those who didn't
Description of pregnancy outcomes | At inclusion
  To describe pregnancy outcomes (gestational diabetis, foetal cardiac rhythm abnormalities, pre-eclampsia/eclampsia, foetal weight abnormalities) of pregnant women who benefited from the intervention with those who didn't, documented from medical file
Description of immediate post-partum outcomes | At inclusion
  To describe immediate post-partum outcomes (vaginal delivery, C-section, post partum bleeding) of pregnant women who benefited from the intervention with those who didn't, documented from medical file
Concentration of micronutrients | At inclusion
  To measure concentration of micronutrients (iron, iodine, zinc, magnesium, vitamins...) of pregnant women
Concentration of heavy metal | At inclusion
  To measure concentration of heavy metal (mercury, lead) of pregnant women
Description of self-esteem | At inclusion
  To describe the self-esteem of pregnant women using the Rosenberg self esteem questionnaire
Description of knowledge of pregnant women on diet | At inclusion
  To describe the level of knowledge on diet of pregant women who benefited from the helath promotion intervention

CONTACTS AND LOCATIONS:
Overall Officials: Celia BASURKO, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Radimer KL, Radimer KL. Measurement of household food security in the USA and other industrialised countries. Public Health Nutr. 2002 Dec;5(6A):859-64. doi: 10.1079/PHN2002385. PMID 12633509
- [Background] Basu S, Meghani A, Siddiqi A. Evaluating the Health Impact of Large-Scale Public Policy Changes: Classical and Novel Approaches. Annu Rev Public Health. 2017 Mar 20;38:351-370. doi: 10.1146/annurev-publhealth-031816-044208. PMID 28384086
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Austin PC. The relative ability of different propensity score methods to balance measured covariates between treated and untreated subjects in observational studies. Med Decis Making. 2009 Nov-Dec;29(6):661-77. doi: 10.1177/0272989X09341755. Epub 2009 Aug 14. PMID 19684288
- See also: Global health in French Guiana : descriptive and comparative study of main health indicators — https://beh.santepubliquefrance.fr/beh/2020/2-3/2020_2-3_1.html
- See also: Mother and child prevention in French Guiana : coping solutions in response to deteriorating living conditions of local populations — https://www.santepubliquefrance.fr/regions/guyane/documents/article/2020/pmi-en-guyane-s-adapter-pour-faire-face-aux-conditions-de-vie-degradees-des-populations-interview
- See also: Heavy metal impregnations in French population. Biosurveillance national program Esteban 2014-2016 — https://www.santepubliquefrance.fr/docs/impregnation-de-la-population-francaise-par-les-metaux-urinaires.-programme-national-de-biosurveillance.-esteban-2014-2016